CLINICAL TRIAL: NCT01554202
Title: Study of the Predictive Markers and the Pathophysiological Mechanisms of Alzheimer's Disease: Transverse and Longitudinal Approach in Anatomical and Functional Multimodal Imaging
Brief Title: Multi-modal Neuroimaging in Alzheimer's Disease
Acronym: IMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A00414-49
Record Dates: First submitted 2012-03-13; First posted 2012-03-14 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; MCI; genetic; AV45-PET
MeSH Terms: conditions — Alzheimer Disease | interventions — Apolipoprotein E4

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Young controls (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Middle age controls (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Elderly controls (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Autosomal dominant forms of early-onset Alzheimer disease (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Subjectif Cognitive Impariment patients (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Mild Cognitive Impairment patients (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Alzheimer Disease patients (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Non degenerative amnsesic syndrome (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Frontotemporal lobe dementia (Experimental): Assessment of memory, circulating tPA dosage, ApoE4, brain imaging examination MRI and PET examinations.
  Interventions: Behavioral: assessment of memory; Biological: circulating tPA dosage; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations

INTERVENTIONS:
Behavioral: assessment of memory
Biological: circulating tPA dosage
Genetic: ApoE4
Other: Brain imaging examination MRI and PET examinations

SUMMARY:
According to estimations, Alzheimer's disease affects approximately 860,000 people aged of more than 65 years in France. This disease is characterized by disorders of cognitive functions, including memory, associated with structural and functional modifications of the brain. These changes are evolving within the pathology progression and can be evaluated with neuropsychological tests (to assess capabilities such as language, orientation, etc.) and also with brain imaging (e.g. MRI). Alzheimer's disease is still poorly understood, nevertheless currently available treatments can slow its development if the disease is diagnosed early enough.

Thus, the objective is to identify markers for early diagnosis of Alzheimer's disease, to better describe the evolution of this disease.

The three main objectives of this project are

* to identify, compare and combine predictive markers of Alzheimer's disease
* to make a significant contribution to the understanding of the pathophysiological mechanisms of Alzheimer's disease
* to study the ability of different neuroimaging techniques to follow the evolution of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Education level > 7 years
* Native language: French
* Medical, neurological, neuropsychological and neuroradiological depth in accordance with the criteria for inclusion and exclusion-specific population, that is to say:

  * Healthy young controls: between 18 and 40 years old; normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.5 SD).
  * Healthy Middle-aged controls: between 40 and 60 years old; without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.5 SD).
  * Healthy Elderly controls: over 60 years old, living at home, without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.5 SD).
  * MCI patients: over 60 years old, presenting the current criteria for amnestic MCI including: i) memory complaint, ii) deficits of the episodic memory (lower performance of at least 1.5 SD from the norm for age and cultural level for one or more scores of episodic memory and iii) normal performances compared to the age and the educational level of all other cognitive functions as memory, including tests to assess cognitive abilities.
  * Alzheimer's patients: presenting the standard criteria of NINCDS-ADRDA probable Alzheimer's disease, including abnormal global cognitive function and deficits in at least two cognitive domains identified by the diagnostic battery and a mild to moderate Alzheimer's disease (MMSE ≥ 15).

Exclusion Criteria:

* The sudden onset of cognitive impairments (as opposed to their slow and gradual installation in Alzheimer's disease)
* A chronic neurological, psychiatric, endocrine, hepatic or infectious complaint
* A history of major disease (an uncontrolled diabetes, a lung, heart, metabolic, hematologic, endocrine disease or a severe cancer);
* A medication that may interfere with memory or metabolic measures
* A alcohol or drugs abuse
* claustrophobia, metallic object in the body
* A predominantly left-hand (score below 50% in Edinburgh Inventory).
* Protected adults, and persons not affiliated with a social security system will not participate in this study.
* The inclusion of a participant in another biomedical research protocol (during the study or within 12 months before inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2008-01; Primary Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of volume change of whole brain, hippocampus and other structural MRI measures | 3 years
Rate of Decline as measured by: Cognitive Tests, Activities of Daily Living, and CDR Sum of Boxes | 3 years
Rates of change on each specified biochemical biomarker | 3 years
Rates of change of glucose metabolism (FDG-PET) | 3 years
Extent of amyloid deposition as measured by 18F-AV45 | 3 years
Group differences for each imaging and biomarker measurement | 3 years
APOE genotype | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de La Sayette, MD, Principal Investigator — University Hospital, Caen
Locations (5):
- France (5):
  - University Hospital Côte de Nacre, Caen
  - University Hospital Roger Salengro, Lille
  - University Hospital Pontchaillou, Rennes
  - University Hospital Rouen, Rouen
  - University Hospital Tours, Tours

REFERENCES:
- [Background] Chetelat G. [Neuroimaging Alzheimer's disease: early diagnosis, monitoring, and mechanism understanding]. Med Sci (Paris). 2011 Feb;27(2):193-8. doi: 10.1051/medsci/2011272193. Epub 2011 Mar 8. French. PMID 21382329
- [Background] Mevel K, Grassiot B, Chetelat G, Defer G, Desgranges B, Eustache F. [The default mode network: cognitive role and pathological disturbances]. Rev Neurol (Paris). 2010 Nov;166(11):859-72. doi: 10.1016/j.neurol.2010.01.008. Epub 2010 Mar 11. French. PMID 20226489
- [Result] La Joie R, Fouquet M, Mezenge F, Landeau B, Villain N, Mevel K, Pelerin A, Eustache F, Desgranges B, Chetelat G. Differential effect of age on hippocampal subfields assessed using a new high-resolution 3T MR sequence. Neuroimage. 2010 Nov 1;53(2):506-14. doi: 10.1016/j.neuroimage.2010.06.024. Epub 2010 Jun 16. PMID 20600996
- [Result] Villain N, Landeau B, Groussard M, Mevel K, Fouquet M, Dayan J, Eustache F, Desgranges B, Chetelat G. A simple way to improve anatomical mapping of functional brain imaging. J Neuroimaging. 2010 Oct;20(4):324-33. doi: 10.1111/j.1552-6569.2010.00470.x. PMID 20331499